CLINICAL TRIAL: NCT01468246
Title: Helping Ourselves, Helping Others: The Young Women's Breast Cancer Study
Brief Title: The Young Women's Breast Cancer Study
Acronym: HOHO
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 06-169
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cohort; Young Women; Survivorship; Fertility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators are collecting blood and tumor specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young Women: Young women with newly diagnosed breast cancer

SUMMARY:
The investigators are conducting a longitudinal cohort study of young women with breast cancer. The investigators identify women age 40 and younger with newly-diagnosed breast cancer from academic and community healthcare institutions. After women consent to the study, they fill-out surveys and give blood samples, and the investigators collect tissue from their breast cancer tumor after it is removed. Women are surveyed every 6 months for the first 3 years after diagnosis, then yearly thereafter for an additional 7 years (for a total follow-up of at least 10 years following diagnosis). The study investigates short and long-term disease and treatment issues, tumor biology and the relationship to patient outcomes, and psychosocial concerns at baseline and in follow-up among a cohort of young women who are newly-diagnosed with breast cancer.

DETAILED DESCRIPTION:
This is a longitudinal cohort study of young women with breast cancer. Over a 6-year period, the investigators aim to identify over 1,600 women age 40 and younger with newly diagnosed breast cancer from academic and community health care institutions. It is anticipated that 1,300 of these women will agree to participate in an observational study. Patient surveys, medical record review, and blood and tissue collection will be utilized. Women will be surveyed every 6 months for the first 3 years after diagnosis, then yearly thereafter for an additional 7 years (for a total follow-up of 10 year following diagnosis). The study will investigate short and long-term disease and treatment issues, and psychosocial concerns at baseline and in follow-up among a cohort of young women (age 40 or younger) newly diagnosed with breast cancer. The investigators aim to characterize the population of young women at diagnosis and in follow-up regarding disease and psychosocial outcomes (e.g., presentation and disease characteristics, treatment patterns and quality of care, short and long-term side effects, and psychosocial concerns including fertility, sexual functioning, and menopausal issues). The investigators will also collect tumor and blood specimens to characterize the tumors, and bank for future studies including molecular evaluations of disease characteristics, genetic variability and hormonal levels in blood. Ultimately, the investigators aim to develop predictors of outcome, and identify areas that may be amenable to intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of breast cancer
* Age 40 or younger at diagnosis
* Informed consent obtained from patient
* Ability to understand written and spoken English to the extent necessary to complete the questionnaires

Exclusion Criteria:

* Inability to understand written and spoken English to the extent necessary to complete the questionnaires
* Absence of informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes women who are newly-diagnosed with breast cancer. They must be 40 or younger at their diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1302 (Actual)
Dates: Start 2006-11; Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Identify a cohort of young women (age 40 or younger) newly diagnosed with breast cancer | 10 years
  Characterize the population of young women at diagnosis and in follow-up regarding disease and psychosocial outcomes (e.g., presentation and disease characteristics including evaluating women with metastatic disease, reported frequency and factors associated with genetic testing, treatment patterns and quality of care, short and long-term side effects, and psychosocial concerns including fertility, sexual functioning, and menopausal issues).
Specimen Collection | 10 years
  Collect tumor and blood specimens to characterize the tumors, and bank for future studies including molecular evaluations of disease characteristics, genetic variability and hormonal levels in blood.

SECONDARY OUTCOMES:
Identify Predictors of Outcome | 10 years
  Ultimately, the investigators aim to develop predictors of outcome and identify areas that may be amenable to intervention for young women with breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Peppercorn, MD, Principal Investigator — Massachusetts General Hospital; Steven Come, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center; Therese Mulvey, MD, Principal Investigator — Mass General/North-Shore Cancer Center; Blair Ardman, MD, Principal Investigator — Lowell General Hospital; Lawrence Blaszkowsky, MD, Principal Investigator — Newton-Wellesley Hospital; Frank G Basile, MD, Principal Investigator — Cape Cod Hospital; Ellen Warner, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Virginia Borges, MD, Principal Investigator — University of Colorado, Denver; Kathryn Ruddy, MD, MPH, Principal Investigator — Mayo Clinic; Katherina Zabicki Calvillo, MD, FACS, Principal Investigator — South Shore Hospital; Jeanna Walsh, MD, Principal Investigator — Dana-Farber/New Hampshire Oncology-Hematology; Natalie Sinclair, MD, Principal Investigator — DF/BWCC at Milford Regional Medical Center
Locations (13):
- United States (12):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - MGH/North Shore Cancer Center, Danvers, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - DF/BWCC at Milford Regional Medical Center, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Collins LC, Marotti JD, Gelber S, Cole K, Ruddy K, Kereakoglow S, Brachtel EF, Schapira L, Come SE, Winer EP, Partridge AH. Pathologic features and molecular phenotype by patient age in a large cohort of young women with breast cancer. Breast Cancer Res Treat. 2012 Feb;131(3):1061-6. doi: 10.1007/s10549-011-1872-9. Epub 2011 Nov 13. PMID 22080245
- [Result] Rosenberg SM, Tamimi RM, Gelber S, Ruddy KJ, Kereakoglow S, Borges VF, Come SE, Schapira L, Winer EP, Partridge AH. Body image in recently diagnosed young women with early breast cancer. Psychooncology. 2013 Aug;22(8):1849-55. doi: 10.1002/pon.3221. Epub 2012 Nov 7. PMID 23132765
- [Result] Rosenberg SM, Tracy MS, Meyer ME, Sepucha K, Gelber S, Hirshfield-Bartek J, Troyan S, Morrow M, Schapira L, Come SE, Winer EP, Partridge AH. Perceptions, knowledge, and satisfaction with contralateral prophylactic mastectomy among young women with breast cancer: a cross-sectional survey. Ann Intern Med. 2013 Sep 17;159(6):373-81. doi: 10.7326/0003-4819-159-6-201309170-00003. PMID 24042365
- [Result] Ruddy KJ, Gelber S, Tamimi RM, Schapira L, Come SE, Meyer ME, Winer EP, Partridge AH. Breast cancer presentation and diagnostic delays in young women. Cancer. 2014 Jan 1;120(1):20-5. doi: 10.1002/cncr.28287. Epub 2013 Nov 11. PMID 24347383
- [Result] Ruddy KJ, Gelber SI, Tamimi RM, Ginsburg ES, Schapira L, Come SE, Borges VF, Meyer ME, Partridge AH. Prospective study of fertility concerns and preservation strategies in young women with breast cancer. J Clin Oncol. 2014 Apr 10;32(11):1151-6. doi: 10.1200/JCO.2013.52.8877. Epub 2014 Feb 24. PMID 24567428
- [Result] Rosenberg SM, Tamimi RM, Gelber S, Ruddy KJ, Bober SL, Kereakoglow S, Borges VF, Come SE, Schapira L, Partridge AH. Treatment-related amenorrhea and sexual functioning in young breast cancer survivors. Cancer. 2014 Aug 1;120(15):2264-71. doi: 10.1002/cncr.28738. Epub 2014 May 28. PMID 24891236
- [Result] Rosenberg SM, Sepucha K, Ruddy KJ, Tamimi RM, Gelber S, Meyer ME, Schapira L, Come SE, Borges VF, Golshan M, Winer EP, Partridge AH. Local Therapy Decision-Making and Contralateral Prophylactic Mastectomy in Young Women with Early-Stage Breast Cancer. Ann Surg Oncol. 2015 Nov;22(12):3809-15. doi: 10.1245/s10434-015-4572-6. Epub 2015 May 1. PMID 25930247
- [Result] Borstelmann NA, Rosenberg SM, Ruddy KJ, Tamimi RM, Gelber S, Schapira L, Come S, Borges V, Morgan E, Partridge AH. Partner support and anxiety in young women with breast cancer. Psychooncology. 2015 Dec;24(12):1679-85. doi: 10.1002/pon.3780. Epub 2015 Mar 13. PMID 25765893
- [Result] Collins LC, Gelber S, Marotti JD, White S, Ruddy K, Brachtel EF, Schapira L, Come SE, Borges VF, Schedin P, Warner E, Wensley T, Tamimi RM, Winer EP, Partridge AH. Molecular Phenotype of Breast Cancer According to Time Since Last Pregnancy in a Large Cohort of Young Women. Oncologist. 2015 Jul;20(7):713-8. doi: 10.1634/theoncologist.2014-0412. Epub 2015 May 29. PMID 26025931
- [Result] Walker HE, Rosenberg SM, Stanton AL, Petrie KJ, Partridge AH. Perceptions, Attributions, and Emotions Toward Endocrine Therapy in Young Women with Breast Cancer. J Adolesc Young Adult Oncol. 2016 Mar;5(1):16-23. doi: 10.1089/jayao.2015.0051. Epub 2015 Dec 17. PMID 26812461
- [Result] Rosenberg SM, Ruddy KJ, Tamimi RM, Gelber S, Schapira L, Come S, Borges VF, Larsen B, Garber JE, Partridge AH. BRCA1 and BRCA2 Mutation Testing in Young Women With Breast Cancer. JAMA Oncol. 2016 Jun 1;2(6):730-6. doi: 10.1001/jamaoncol.2015.5941. PMID 26867710
- [Result] Goddard ET, Hill RC, Nemkov T, D'Alessandro A, Hansen KC, Maller O, Mongoue-Tchokote S, Mori M, Partridge AH, Borges VF, Schedin P. The Rodent Liver Undergoes Weaning-Induced Involution and Supports Breast Cancer Metastasis. Cancer Discov. 2017 Feb;7(2):177-187. doi: 10.1158/2159-8290.CD-16-0822. Epub 2016 Dec 14. PMID 27974414
- [Result] Olsen SN, Wronski A, Castano Z, Dake B, Malone C, De Raedt T, Enos M, DeRose YS, Zhou W, Guerra S, Loda M, Welm A, Partridge AH, McAllister SS, Kuperwasser C, Cichowski K. Loss of RasGAP Tumor Suppressors Underlies the Aggressive Nature of Luminal B Breast Cancers. Cancer Discov. 2017 Feb;7(2):202-217. doi: 10.1158/2159-8290.CD-16-0520. Epub 2016 Dec 14. PMID 27974415
- [Result] Park EM, Gelber S, Rosenberg SM, Seah DSE, Schapira L, Come SE, Partridge AH. Anxiety and Depression in Young Women With Metastatic Breast Cancer: A Cross-Sectional Study. Psychosomatics. 2018 May-Jun;59(3):251-258. doi: 10.1016/j.psym.2018.01.007. Epub 2018 Jan 31. PMID 29525523
- [Result] von Hippel C, Rosenberg SM, Austin SB, Sprunck-Harrild K, Ruddy KJ, Schapira L, Come S, Borges VF, Partridge AH. Identifying distinct trajectories of change in young breast cancer survivors' sexual functioning. Psychooncology. 2019 May;28(5):1033-1040. doi: 10.1002/pon.5047. Epub 2019 Mar 13. PMID 30817075
- [Result] Wassermann J, Gelber SI, Rosenberg SM, Ruddy KJ, Tamimi RM, Schapira L, Borges VF, Come SE, Meyer ME, Partridge AH. Nonadherent behaviors among young women on adjuvant endocrine therapy for breast cancer. Cancer. 2019 Sep 15;125(18):3266-3274. doi: 10.1002/cncr.32192. Epub 2019 May 23. PMID 31120571
- [Result] Rath M, Li Q, Li H, Lindstrom S, Miron A, Miron P, Dowton AE, Meyer ME, Larson BG, Pomerantz M, Seo JH, Collins LC, Vardeh H, Brachtel E, Come SE, Borges V, Schapira L, Tamimi RM, Partridge AH, Freedman M, Ruddy KJ. Evaluation of significant genome-wide association studies risk - SNPs in young breast cancer patients. PLoS One. 2019 May 24;14(5):e0216997. doi: 10.1371/journal.pone.0216997. eCollection 2019. PMID 31125336
- [Result] Rosenberg SM, Vaz-Luis I, Gong J, Rajagopal PS, Ruddy KJ, Tamimi RM, Schapira L, Come S, Borges V, de Moor JS, Partridge AH. Employment trends in young women following a breast cancer diagnosis. Breast Cancer Res Treat. 2019 Aug;177(1):207-214. doi: 10.1007/s10549-019-05293-x. Epub 2019 May 30. PMID 31147983
- [Result] Lee GE, Rosenberg SM, Mayer EL, Borges V, Meyer ME, Schapira L, Come SE, Partridge AH. Contemporary management of breast cancer during pregnancy and subsequent lactation in a multicenter cohort of young women with breast cancer. Breast J. 2019 Nov;25(6):1104-1110. doi: 10.1111/tbj.13431. Epub 2019 Jul 18. PMID 31318125
- [Result] Poorvu PD, Gelber SI, Rosenberg SM, Ruddy KJ, Tamimi RM, Collins LC, Peppercorn J, Schapira L, Borges VF, Come SE, Warner E, Jakubowski DM, Russell C, Winer EP, Partridge AH. Prognostic Impact of the 21-Gene Recurrence Score Assay Among Young Women With Node-Negative and Node-Positive ER-Positive/HER2-Negative Breast Cancer. J Clin Oncol. 2020 Mar 1;38(7):725-733. doi: 10.1200/JCO.19.01959. Epub 2019 Dec 6. PMID 31809240
- [Result] Pak LM, Gaither R, Rosenberg SM, Ruddy KJ, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Warner E, Snow C, Collins LC, King TA, Partridge AH. Tumor phenotype and concordance in synchronous bilateral breast cancer in young women. Breast Cancer Res Treat. 2021 Apr;186(3):815-821. doi: 10.1007/s10549-020-06027-0. Epub 2020 Nov 26. PMID 33242164
- [Result] Parsons HA, Rhoades J, Reed SC, Gydush G, Ram P, Exman P, Xiong K, Lo CC, Li T, Fleharty M, Kirkner GJ, Rotem D, Cohen O, Yu F, Fitarelli-Kiehl M, Leong KW, Hughes ME, Rosenberg SM, Collins LC, Miller KD, Blumenstiel B, Trippa L, Cibulskis C, Neuberg DS, DeFelice M, Freeman SS, Lennon NJ, Wagle N, Ha G, Stover DG, Choudhury AD, Getz G, Winer EP, Meyerson M, Lin NU, Krop I, Love JC, Makrigiorgos GM, Partridge AH, Mayer EL, Golub TR, Adalsteinsson VA. Sensitive Detection of Minimal Residual Disease in Patients Treated for Early-Stage Breast Cancer. Clin Cancer Res. 2020 Jun 1;26(11):2556-2564. doi: 10.1158/1078-0432.CCR-19-3005. Epub 2020 Mar 13. PMID 32170028
- [Result] Vazquez D, Rosenberg S, Gelber S, Ruddy KJ, Morgan E, Recklitis C, Come S, Schapira L, Partridge AH. Posttraumatic stress in breast cancer survivors diagnosed at a young age. Psychooncology. 2020 Aug;29(8):1312-1320. doi: 10.1002/pon.5438. Epub 2020 Jul 9. PMID 32515073
- [Result] Rosenberg SM, Dominici LS, Gelber S, Poorvu PD, Ruddy KJ, Wong JS, Tamimi RM, Schapira L, Come S, Peppercorn JM, Borges VF, Partridge AH. Association of Breast Cancer Surgery With Quality of Life and Psychosocial Well-being in Young Breast Cancer Survivors. JAMA Surg. 2020 Nov 1;155(11):1035-1042. doi: 10.1001/jamasurg.2020.3325. PMID 32936216
- [Result] Borstelmann NA, Rosenberg S, Gelber S, Zheng Y, Meyer M, Ruddy KJ, Schapira L, Come S, Borges V, Cadet T, Maramaldi P, Partridge AH. Partners of young breast cancer survivors: a cross-sectional evaluation of psychosocial concerns, coping, and mental health. J Psychosoc Oncol. 2020 Nov-Dec;38(6):670-686. doi: 10.1080/07347332.2020.1823546. Epub 2020 Oct 1. PMID 33000705
- [Result] Poorvu PD, Gelber SI, Zheng Y, Ruddy KJ, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Lambertini M, Rosenberg SM, Partridge AH. Pregnancy after breast cancer: Results from a prospective cohort of young women with breast cancer. Cancer. 2021 Apr 1;127(7):1021-1028. doi: 10.1002/cncr.33342. Epub 2020 Dec 1. PMID 33259061
- [Result] Lambertini M, Ameye L, Hamy AS, Zingarello A, Poorvu PD, Carrasco E, Grinshpun A, Han S, Rousset-Jablonski C, Ferrari A, Paluch-Shimon S, Cortesi L, Senechal C, Miolo G, Pogoda K, Perez-Fidalgo JA, De Marchis L, Ponzone R, Livraghi L, Estevez-Diz MDP, Villarreal-Garza C, Dieci MV, Clatot F, Berliere M, Graffeo R, Teixeira L, Cordoba O, Sonnenblick A, Luna Pais H, Ignatiadis M, Paesmans M, Partridge AH, Caron O, Saule C, Del Mastro L, Peccatori FA, Azim HA Jr. Pregnancy After Breast Cancer in Patients With Germline BRCA Mutations. J Clin Oncol. 2020 Sep 10;38(26):3012-3023. doi: 10.1200/JCO.19.02399. Epub 2020 Jul 16. PMID 32673153
- [Result] Sella T, Gelber SI, Poorvu PD, Kim HJ, Dominici L, Guzman-Arocho YD, Collins L, Ruddy KJ, Tamimi RM, Peppercorn JM, Schapira L, Borges VF, Come SE, Warner E, Snow C, Jakubowski DM, Russell CA, Winer EP, Rosenberg SM, Partridge AH. Response to neoadjuvant chemotherapy and the 21-gene Breast Recurrence Score test in young women with estrogen receptor-positive early breast cancer. Breast Cancer Res Treat. 2021 Feb;186(1):157-165. doi: 10.1007/s10549-020-05989-5. Epub 2020 Nov 4. PMID 33150547
- [Result] Kim HJ, Dominici L, Rosenberg SM, Zheng Y, Pak LM, Poorvu PD, Ruddy KJ, Tamimi R, Schapira L, Come SE, Peppercorn J, Borges VF, Warner E, Vardeh H, Collins LC, Gaither R, King TA, Partridge AH. Surgical Treatment After Neoadjuvant Systemic Therapy in Young Women With Breast Cancer: Results From a Prospective Cohort Study. Ann Surg. 2022 Jul 1;276(1):173-179. doi: 10.1097/SLA.0000000000004296. Epub 2020 Dec 23. PMID 33378304
- [Result] Sella T, Poorvu PD, Ruddy KJ, Gelber SI, Tamimi RM, Peppercorn JM, Schapira L, Borges VF, Come SE, Partridge AH, Rosenberg SM. Impact of fertility concerns on endocrine therapy decisions in young breast cancer survivors. Cancer. 2021 Aug 15;127(16):2888-2894. doi: 10.1002/cncr.33596. Epub 2021 Apr 22. PMID 33886123
- [Result] Kuijer A, Dominici LS, Rosenberg SM, Hu J, Gelber S, Di Lascio S, Wong JS, Ruddy KJ, Tamimi RM, Schapira L, Borges VF, Come SE, Sprunck-Harrild K, Partridge AH, King TA. Arm Morbidity After Local Therapy for Young Breast Cancer Patients. Ann Surg Oncol. 2021 Oct;28(11):6071-6082. doi: 10.1245/s10434-021-09947-3. Epub 2021 Apr 21. PMID 33881656
- [Result] Guzman-Arocho YD, Rosenberg SM, Garber JE, Vardeh H, Poorvu PD, Ruddy KJ, Kirkner G, Snow C, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Brachtel EF, Marotti JD, Warner E, Partridge AH, Collins LC. Clinicopathological features and BRCA1 and BRCA2 mutation status in a prospective cohort of young women with breast cancer. Br J Cancer. 2022 Feb;126(2):302-309. doi: 10.1038/s41416-021-01597-2. Epub 2021 Oct 26. PMID 34703009
- [Result] Schapira L, Zheng Y, Gelber SI, Poorvu P, Ruddy KJ, Tamimi RM, Peppercorn J, Come SE, Borges VF, Partridge AH, Rosenberg SM. Trajectories of fear of cancer recurrence in young breast cancer survivors. Cancer. 2022 Jan 15;128(2):335-343. doi: 10.1002/cncr.33921. Epub 2021 Oct 6. PMID 34614212
- [Result] Dominici L, Hu J, Zheng Y, Kim HJ, King TA, Ruddy KJ, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Warner E, Wong JS, Partridge AH, Rosenberg SM. Association of Local Therapy With Quality-of-Life Outcomes in Young Women With Breast Cancer. JAMA Surg. 2021 Oct 1;156(10):e213758. doi: 10.1001/jamasurg.2021.3758. Epub 2021 Oct 13. PMID 34468718
- [Result] Lambertini M, Blondeaux E, Bruzzone M, Perachino M, Anderson RA, de Azambuja E, Poorvu PD, Kim HJ, Villarreal-Garza C, Pistilli B, Vaz-Luis I, Saura C, Ruddy KJ, Franzoi MA, Sertoli C, Ceppi M, Azim HA Jr, Amant F, Demeestere I, Del Mastro L, Partridge AH, Pagani O, Peccatori FA. Pregnancy After Breast Cancer: A Systematic Review and Meta-Analysis. J Clin Oncol. 2021 Oct 10;39(29):3293-3305. doi: 10.1200/JCO.21.00535. Epub 2021 Jul 1. PMID 34197218
- [Result] Poorvu PD, Hu J, Zheng Y, Gelber SI, Ruddy KJ, Tamimi RM, Peppercorn JM, Schapira L, Borges VF, Come SE, Warner E, Lambertini M, Rosenberg SM, Partridge AH. Treatment-related amenorrhea in a modern, prospective cohort study of young women with breast cancer. NPJ Breast Cancer. 2021 Jul 27;7(1):99. doi: 10.1038/s41523-021-00307-8. PMID 34315890
- [Result] Lambertini M, Ceppi M, Hamy AS, Caron O, Poorvu PD, Carrasco E, Grinshpun A, Punie K, Rousset-Jablonski C, Ferrari A, Paluch-Shimon S, Toss A, Senechal C, Puglisi F, Pogoda K, Perez-Fidalgo JA, De Marchis L, Ponzone R, Livraghi L, Estevez-Diz MDP, Villarreal-Garza C, Dieci MV, Clatot F, Duhoux FP, Graffeo R, Teixeira L, Cordoba O, Sonnenblick A, Ferreira AR, Partridge AH, Di Meglio A, Saule C, Peccatori FA, Bruzzone M, t'Kint de Roodenbeke MD, Ameye L, Balmana J, Del Mastro L, Azim HA Jr. Clinical behavior and outcomes of breast cancer in young women with germline BRCA pathogenic variants. NPJ Breast Cancer. 2021 Feb 12;7(1):16. doi: 10.1038/s41523-021-00224-w. PMID 33579978
- [Result] Borstelmann NA, Gray TF, Gelber S, Rosenberg S, Zheng Y, Meyer M, Ruddy KJ, Schapira L, Come S, Borges V, Cadet T, Maramaldi P, Partridge AH. Psychosocial issues and quality of life of parenting partners of young women with breast cancer. Support Care Cancer. 2022 May;30(5):4265-4274. doi: 10.1007/s00520-022-06852-7. Epub 2022 Jan 28. PMID 35091846
- [Result] Sella T, Ruddy KJ, Carey LA, Partridge AH. Optimal Endocrine Therapy in Premenopausal Women: A Pragmatic Approach to Unanswered Questions. JCO Oncol Pract. 2022 Mar;18(3):211-216. doi: 10.1200/OP.21.00482. Epub 2021 Oct 12. PMID 34637342
- [Result] Krasne M, Ruddy KJ, Poorvu PD, Gelber SI, Tamimi RM, Schapira L, Peppercorn J, Come SE, Borges VF, Partridge AH, Rosenberg SM. Coping strategies and anxiety in young breast cancer survivors. Support Care Cancer. 2022 Nov;30(11):9109-9116. doi: 10.1007/s00520-022-07325-7. Epub 2022 Aug 20. PMID 35986100
- [Result] Lewinsohn R, Zheng Y, Rosenberg SM, Ruddy KJ, Tamimi RM, Schapira L, Peppercorn J, Borges VF, Come S, Snow C, Ginsburg ES, Partridge AH. Fertility Preferences and Practices Among Young Women With Breast Cancer: Germline Genetic Carriers Versus Noncarriers. Clin Breast Cancer. 2023 Apr;23(3):317-323. doi: 10.1016/j.clbc.2022.12.012. Epub 2022 Dec 22. PMID 36628811
- [Result] Rosenberg SM, Zheng Y, Gelber S, Ruddy KJ, Poorvu P, Sella T, Tamimi RM, Wassermann J, Schapira L, Borges VF, Come S, Peppercorn J, Sepucha KR, Partridge AH. Adjuvant endocrine therapy non-initiation and non-persistence in young women with early-stage breast cancer. Breast Cancer Res Treat. 2023 Feb;197(3):547-558. doi: 10.1007/s10549-022-06810-1. Epub 2022 Nov 27. PMID 36436128
- [Result] Sella T, Zheng Y, Tan-Wasielewski Z, Rosenberg SM, Poorvu PD, Tayob N, Ruddy KJ, Gelber SI, Tamimi RM, Schapira L, Come SE, Peppercorn JM, Borges VF, Partridge AH, Ligibel JA. Body weight changes and associated predictors in a prospective cohort of young breast cancer survivors. Cancer. 2022 Sep 1;128(17):3158-3169. doi: 10.1002/cncr.34342. Epub 2022 Jul 1. PMID 35775874
- [Result] Sella T, Fell GG, Miller PG, Gibson CJ, Rosenberg SM, Snow C, Stover DG, Ruddy KJ, Peppercorn JM, Schapira L, Borges VF, Come SE, Warner E, Frank E, Neuberg DS, Ebert BL, Partridge AH. Patient perspectives on testing for clonal hematopoiesis of indeterminate potential. Blood Adv. 2022 Dec 27;6(24):6151-6161. doi: 10.1182/bloodadvances.2022008376. PMID 36129839
- [Result] Tesch ME, Rosenberg SM, Collins LC, Wong JS, Dominici L, Ruddy KJ, Tamimi R, Schapira L, Borges VF, Warner E, Come SE, Partridge AH. Clinicopathologic Features, Treatment Patterns, and Disease Outcomes in a Modern, Prospective Cohort of Young Women Diagnosed with Ductal Carcinoma In Situ. Ann Surg Oncol. 2022 Dec;29(13):8048-8057. doi: 10.1245/s10434-022-12361-y. Epub 2022 Aug 12. PMID 35960452
- [Result] Waks AG, Kim D, Jain E, Snow C, Kirkner GJ, Rosenberg SM, Oh C, Poorvu PD, Ruddy KJ, Tamimi RM, Peppercorn J, Schapira L, Borges VF, Come SE, Brachtel EF, Warner E, Collins LC, Partridge AH, Wagle N. Somatic and Germline Genomic Alterations in Very Young Women with Breast Cancer. Clin Cancer Res. 2022 Jun 1;28(11):2339-2348. doi: 10.1158/1078-0432.CCR-21-2572. PMID 35101884
- [Derived] Singh MP, Gupta S, Singh M, Ambrish C, Kurmi P, Gangwani DK, Naganna J, Sethuraman R, Dhumal V, Behera S, Patel PM, Patil DM, Lakhwani LK, Ghadge PS, Mehta SC, Joglekar SJ. Efficacy and Safety of Triple Fixed Dose Combination of Dapagliflozin + Sitagliptin + Metformin IR in Indian Patients with Type 2 Diabetes Mellitus: A Randomized, Phase 3 Study in Comparison with Dual FDC Sitagliptin + Metformin IR. Adv Ther. 2025 Oct;42(10):5187-5201. doi: 10.1007/s12325-025-03323-3. Epub 2025 Aug 19. PMID 40828352
- [Derived] Rosenberg SM, Zheng Y, Ruddy K, Poorvu PD, Snow C, Kirkner GJ, Meyer ME, Tamimi RM, Schapira L, Peppercorn J, Come S, Borges VF, Warner E, Gelber S, Collins L, Winer EP, Partridge AH. Helping ourselves, helping others: the Young Women's Breast Cancer Study (YWS) - a multisite prospective cohort study to advance the understanding of breast cancer diagnosed in women aged 40 years and younger. BMJ Open. 2024 Jul 1;14(6):e081157. doi: 10.1136/bmjopen-2023-081157. PMID 38951008